CLINICAL TRIAL: NCT01959256
Title: Visual Perceptual Learning for the Treatment of Visual Field Defect
Acronym: VIVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dong-Wha Kang, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIVID
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Stroke; Visual Field Defect
Keywords: Stroke; Visual Field Defect; Visual perceptual learning; Brain connectivity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Learning (Experimental): Visual perceptual learning (VPL) group
  Interventions: Behavioral: Visual perceptual learning
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Visual perceptual learning — 24 times of training for visual perceptual learning
  Arms: Learning

SUMMARY:
This study will test the hypothesis whether visual field defect caused by chronic stroke could be improved by visual perceptual learning. The secondary hypothesis is that improvement of visual field defect would be accompanied by connectivity changes in visual networks. In addition, investigators will evaluate whether improvement of visual field defect could achieve improvement of subjective visual function.

DETAILED DESCRIPTION:
Study design: A PROBE (Prospective, Randomized, Open-label, Blinded-endpoint) design

Methods:

1. Visual perceptual learning (VPL) group

   1. Visual perceptual learning (24 times for 2 months, 3 times per week) in visual field defect areas
   2. At baseline and post-VPL evaluations (2 months after): Structural & Functional MRIs, Visual field tests, Visual evoked potential, Visual cognitive tests, Subjective visual function questionnaires
2. Control group

   1. At baseline and 2-months later: No VPL, Structural & Functional MRIs, Visual field tests, Visual evoked potential, Visual cognitive tests, Subjective visual function questionnaires
   2. Visual perceptual learning after 2-month follow-up evaluation (24 times for 2 months, 3 times per week)

   (The patients who were stratified by age (over 65 years old or not) and degree of visual field defect (quadrantanopia or complete hemianopia) will be randomly assigned into the learning and control group.)
3. Investigations

   1. Improvement of visual field test scores between VPL group and control group
   2. Analysis of brain network changes in MRI data
   3. Correlation analysis of improvement of visual field defect and MRI data
   4. Correlation analysis of improvement of visual field defect and visual evoked potential (VEP) data
   5. Correlation analysis of improvement of visual field defect and neuropsychological data

ELIGIBILITY:
Inclusion Criteria:

1. The patient has chronic stroke more than 6 months after onset.
2. The patient has visual field defect (Quadrantanopia or Hemianopia).
3. The patient has corrected eyesight 0.7 or above.

Exclusion Criteria:

1. The patient has contraindication to MRI scan.
2. The patient has cognitive impairment (Mini-Mental Status Exam score <24).
3. The patient has ophthalmologic diseases (e.g., glaucoma, cataract).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Improvement of visual field scores in visual field defect areas | At 2 months (plus or minus 7 days) after baseline evaluation
  Improvement of mean deviation scores in defected areas by Humphrey 750i Field test

SECONDARY OUTCOMES:
Performance of visual perceptual learning | At 2 months (plus or minus 7 days) after baseline evaulation
  Performance (scores) of visual perceptual learning
Connectivity changes in MRI | Between baseline and 2 months (plus or minus 7 days) after
  1. Functional connectivity changes in resting-state functional MRI
  2. Structural connectivity changes in diffusion tensor imaging
Improvement of visual field score in whole visual field area | At 2 months (plus or minus 7days) after baseline evaluation
  Improvement of mean deviation scores in whole visual field by Humphrey 750i Field test
Change of subjective visual function | At 2 months (plus or minus 7days) after baseline evaluation
  1. Change in Korean version of National Eye institute Visual Functioning Questionnaire-25 (NEI-VFQ-25)
  2. Change of subjective visual field area
Changes of visual evoked potential | Between baseline and 2 months (plus or minus 7 days) after
  Changes between baseline and 2 months after in half-field visual evoked potential (VEP) data

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wha Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea